CLINICAL TRIAL: NCT06619158
Title: Long-term Effectiveness of Zirconia Glaze Removal and Polish As an Adjunct to Non-surgical Therapy in Treatment of Persistent Peri-implant Mucositis
Brief Title: Effectiveness of Zirconia Glaze Removal and Polish in the Treatment of Peri-implant Mucositis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Chrysi Stavropoulou, Assistant professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H2024:048
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Peri-Implantitis and Peri-implant Mucositis
Keywords: zirconia glaze removal, crown modification
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Crown modification with glaze removal and polish of implant crown
  Interventions: Procedure: Crown modification
- Group B (No Intervention): No intervention will be applied. The crown will be removed and superficially cleaned

INTERVENTIONS:
Procedure: Crown modification — Zirconia glaze removal and polish after crown removal to reduce roughness and prohibit plaque adhesion
  Arms: Group A

SUMMARY:
This clinical trial is being conducted to study peri-implant mucositis (inflammation in the gums around dental implant that does not extend into the implant-supporting bone). There are currently no available treatment options able to provide long-term resolution of implant gum inflammation even with our current gold standard treatment of non-surgical cleanings and oral hygiene instructions. The purpose of the study is to compare the effect of crown glaze removal and subsequent polishing in addition to mechanical debridement compared to only mechanical debridement on the implant affected by implant gum inflammation.

In this study, participants will be randomized (put into a group by chance) into one of 2 study groups, groups A and B.

Group A: The implant crown will be cleaned with titanium scaling instruments and powered instruments. The screw-retained crown will be removed and the remaining build-up on the crown will be photographed. The crown will then be sent to a lab technician who will remove the glaze and polish the crown only in the areas that sit under the gums.

Group B: The implant crown will be cleaned with titanium scaling instruments and powered instruments. The screw-retained crown will be removed and the remaining build-up on the crown will be photographed. The crown will then be sent to a lab technician to perform a superficial cleaning only.

In both groups, the crown will be placed back on the implant and customized oral hygiene instructions will be provided.

The study will require four appointment. Appointment #1 is the screening appointment and will take 30-60 minutes. Appointment #2 is when treatment is delivered and will occur within 4 weeks of appointment #1. Appointment #3 is for the short-term follow-up and will occur within 60-70 days of appointment #2. Appointment #4 is for the long-term follow-up and will occur within 12-13 months of appointment #2. All these appointment will be in an outpatient setting at the institutional graduate periodontics clinic.

A total of 2 x-rays will be taken of the implant. One will be taken during appointment #1 to assess the bone around the implant. One will be taken during appointment #2 to ensure that the crown is fully seated when the crown is re-inserted.

The following information will be collected in appointment #1: gum measurements around the implants, how tight the implant contacts adjacent teeth, when the crown was delivered, previous cleanings around the implant, age, sex, gender, previous systemic antibiotic use in the last 2 weeks, smoking habits, presence of diabetes and HbA1C values.

At appointments #2, 3, and 4, the following information will be collected: plaque around implant, gum measurements around implants, previous systemic antibiotic use in the last 2 weeks, smoking habits, presence of diabetes and HbA1C values, gum fluid samples around the implant crown. In appointment #4, additionally, information on how the implant has been cleaned throughout the year will be collected.

DETAILED DESCRIPTION:
The study's objectives are:

1. To determine whether a smooth crown surface (<0.2 μm Ra) can be established in-vitro after glaze removal and polishing based on adapted protocol from Go et al., 2019.
2. To determine the effectiveness of submucosal non-surgical hand and powered instrumentation in removal of plaque and calculus.
3. To assess the short- and long-term effectiveness of submucosal zirconia glaze removal and polishing as an adjunct to non-surgical therapy for treatment of persistent peri-implant mucositis. The null hypothesis is that the polishing protocol will not produce any significant differences in the resolution of inflammation compared to crown removal as part of the non-surgical debridement.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 single screw-retained zirconia glazed implant crown which is in function for at least 1 year, with adequate contact points, submucosal crown margins, no adjacent implants, adequate keratinized tissue (2mm or more), and peri-implant mucositis that persists despite recent (within the past 6 months) non-surgical debridement

Exclusion Criteria:

* Contraindications to routine dental treatment Open interproximal contacts, splinted implant prosthesis, peri-implant health, peri-implantitis, cemented crown , removable implant prosthesis, recession past the implant platform Systemic antibiotic use within the last 2 weeks heavy smokers (more than 10 cigarettes/day) uncontrolled diabetes (HbA1C more than 7.0%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
mBI long term | 12 months following treatment
  modified Bleeding index (mBI) around the implant long term (12 months following treatment)
mBI short term | 60-70 days following treatment
  modified bleeding index (mBI) around the implant short term (60-70 days following treatment)
residual plaque and calculus | baseline
  % of plaque and calculus on the subgingival surface of crown

SECONDARY OUTCOMES:
PI long term | 12 months following treatment
  plaque index (PI) around implant long term
PD short term | 60-70 days following treatment
  probing depth (PD) around implant short term
PD long term | 12 months following treatment
  probing depth (PD) around implant long term
PI short term | 60-70 days following treatment
  plaque index (PI) around implant short term
IL-1β baseline | baseline
  level of IL-1β in the peri-implant crevicular fluid
IL-1β short-term | 60-70 days following treatment
  level of IL-1β in the peri-implant crevicular fluid
IL-1β long-term | 12 months following treatment
  level of IL-1β in the peri-implant crevicular fluid
INF-γ baseline | baseline
  level of INF-γ in the peri-implant crevicular fluid
INF-γ short-term | 60-70 days following treatment
  level of INF-γ in the peri-implant crevicular fluid
INF-γ long-term | 12 months following treatment
  level of INF-γ in the peri-implant crevicular fluid
IL-2 baseline | baseline
  level of IL-2 in peri-implant crevicular fluid
IL-2 short-term | 60-70 days following treatment
  level of IL-2 in the peri-implant crevicular fluid
IL-2 long-term | 12 months following treatment
  level of IL-2 in the peri-implant crevicular fluid
IL-4 baseline | baseline
  level of IL-4 in the peri-implant crevicular fluid
IL-4 short-term | 60-70 days following treatment
  level of peri-implant crevicular fluid
IL-4 long-term | 12 months following treatment
  level of IL-4 in the peri-implant crevicular fluid
IL-6 baseline | baseline
  level of IL-6 in peri-implant crevicular fluid
IL-6 short-term | 60-70 days following treatment
  level of IL-6 in peri-implant crevicular fluid
Il-6 long-term | 12 months following treatment
  level of IL-6 in the peri-implant crevicular fluid
IL-8 baseline | baseline
  level of IL-8 in peri-implant crevicular fluid
IL-8 short-term | 60-70 days following treatment
  level of IL-8 in peri-implant crevicular fluid
IL-8 long-term | 12 months following treatment
  level of IL-8 in peri-implant crevicular fluid
IL-10 baseline | baseline
  level of IL-10 in peri-implant crevicular fluid
IL-10 short term | 60-70 days following treatment
  level of IL-10 in peri-implant crevicular fluid
IL-10 long-term | 12 months following treatment
  level of IL-10 in peri-implant crevicular fluid
TNF-α baseline | baseline
  level of TNF-α in peri-implant crevicular fluid
TNF-α short-term | 60-70 days following treatment
  level of TNF-α in peri-implant crevicular fluid
TNF-α long-term | 12 months following treatment
  level of TNF-α in the peri-implant crevicular fluid

CONTACTS AND LOCATIONS:
Overall Officials: Chrysi Stavropoulou, DDS, MDent(Perio), Principal Investigator — University of Manitoba
Locations (1):
- Dr Sam Borden Periodontology Specialty Clinic, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yu P, Wang C, Zhou J, Jiang L, Xue J, Li W. Influence of Surface Properties on Adhesion Forces and Attachment of Streptococcus mutans to Zirconia In Vitro. Biomed Res Int. 2016;2016:8901253. doi: 10.1155/2016/8901253. Epub 2016 Nov 15. PMID 27975061
- [Background] Tete S, Zizzari VL, Borelli B, De Colli M, Zara S, Sorrentino R, Scarano A, Gherlone E, Cataldi A, Zarone F. Proliferation and adhesion capability of human gingival fibroblasts onto zirconia, lithium disilicate and feldspathic veneering ceramic in vitro. Dent Mater J. 2014;33(1):7-15. doi: 10.4012/dmj.2013-185. PMID 24492105
- [Background] Tajti P, Solyom E, Czumbel LM, Szabo B, Fazekas R, Nemeth O, Hermann P, Gerber G, Hegyi P, Mikulas K. Monolithic zirconia as a valid alternative to metal-ceramic for implant-supported single crowns in the posterior region: A systematic review and meta-analysis of randomized controlled trials. J Prosthet Dent. 2024 Nov;132(5):881-889. doi: 10.1016/j.prosdent.2023.05.006. Epub 2023 Jun 21. PMID 37349158
- [Background] Sirinirund B, Siqueira R, Li J, Mendonca G, Zalucha J, Wang HL. Effects of crown contour on artificial biofilm removal efficacy with interdental cleaning aids: An in vitro study. Clin Oral Implants Res. 2023 Aug;34(8):783-792. doi: 10.1111/clr.14105. Epub 2023 Jun 3. PMID 37269176
- [Background] Scotti R, Zanini Kantorski K, Scotti N, Monaco C, Valandro LF, Bottino MA. Early biofilm colonization on polished- and glazed-zirconium ceramic surface. Preliminary results. Minerva Stomatol. 2006 Sep;55(9):493-502. English, Italian. PMID 17146428
- [Background] Renvert S, Hirooka H, Polyzois I, Kelekis-Cholakis A, Wang HL; Working Group 3. Diagnosis and non-surgical treatment of peri-implant diseases and maintenance care of patients with dental implants - Consensus report of working group 3. Int Dent J. 2019 Sep;69(Suppl 2):12-17. doi: 10.1111/idj.12490. PMID 31478575
- [Background] Priest G. A Current Perspective on Screw-Retained Single-Implant Restorations: A Review of Pertinent Literature. J Esthet Restor Dent. 2017 May 6;29(3):161-171. doi: 10.1111/jerd.12283. Epub 2017 Jan 23. PMID 28112854
- [Background] Mombelli A, van Oosten MA, Schurch E Jr, Land NP. The microbiota associated with successful or failing osseointegrated titanium implants. Oral Microbiol Immunol. 1987 Dec;2(4):145-51. doi: 10.1111/j.1399-302x.1987.tb00298.x. No abstract available. PMID 3507627
- [Background] Menezes KM, Fernandes-Costa AN, Silva-Neto RD, Calderon PS, Gurgel BC. Efficacy of 0.12% Chlorhexidine Gluconate for Non-Surgical Treatment of Peri-Implant Mucositis. J Periodontol. 2016 Nov;87(11):1305-1313. doi: 10.1902/jop.2016.160144. Epub 2016 Jul 8. PMID 27389963
- [Background] Lee CT, Huang YW, Zhu L, Weltman R. Prevalences of peri-implantitis and peri-implant mucositis: systematic review and meta-analysis. J Dent. 2017 Jul;62:1-12. doi: 10.1016/j.jdent.2017.04.011. Epub 2017 May 3. PMID 28478213
- [Background] Kim W, Li XC, Bidra AS. Clinical outcomes of implant-supported monolithic zirconia crowns and fixed partial dentures: A systematic review. J Prosthodont. 2023 Feb;32(2):102-107. doi: 10.1111/jopr.13575. Epub 2022 Aug 18. PMID 35929416
- [Background] Katafuchi M, Weinstein BF, Leroux BG, Chen YW, Daubert DM. Restoration contour is a risk indicator for peri-implantitis: A cross-sectional radiographic analysis. J Clin Periodontol. 2018 Feb;45(2):225-232. doi: 10.1111/jcpe.12829. Epub 2017 Dec 5. PMID 28985447
- [Background] Jepsen S, Berglundh T, Genco R, Aass AM, Demirel K, Derks J, Figuero E, Giovannoli JL, Goldstein M, Lambert F, Ortiz-Vigon A, Polyzois I, Salvi GE, Schwarz F, Serino G, Tomasi C, Zitzmann NU. Primary prevention of peri-implantitis: managing peri-implant mucositis. J Clin Periodontol. 2015 Apr;42 Suppl 16:S152-7. doi: 10.1111/jcpe.12369. PMID 25626479
- [Background] Heitz-Mayfield LJ, Salvi GE, Botticelli D, Mombelli A, Faddy M, Lang NP; Implant Complication Research Group. Anti-infective treatment of peri-implant mucositis: a randomised controlled clinical trial. Clin Oral Implants Res. 2011 Mar;22(3):237-41. doi: 10.1111/j.1600-0501.2010.02078.x. Epub 2011 Jan 20. PMID 21251076
- [Background] Hallstrom H, Persson GR, Lindgren S, Olofsson M, Renvert S. Systemic antibiotics and debridement of peri-implant mucositis. A randomized clinical trial. J Clin Periodontol. 2012 Jun;39(6):574-81. doi: 10.1111/j.1600-051X.2012.01884.x. PMID 22571225
- [Background] Go H, Park H, Lee J, Seo H, Lee S. Effect of various polishing burs on surface roughness and bacterial adhesion in pediatric zirconia crowns. Dent Mater J. 2019 Mar 31;38(2):311-316. doi: 10.4012/dmj.2018-106. Epub 2019 Feb 28. PMID 30814454
- [Background] Eickholz P, Grotkamp FL, Steveling H, Muhling J, Staehle HJ. Reproducibility of peri-implant probing using a force-controlled probe. Clin Oral Implants Res. 2001 Apr;12(2):153-8. doi: 10.1034/j.1600-0501.2001.012002153.x. PMID 11251665
- [Background] Dommisch H, Hoedke D, Valles C, Vilarrasa J, Jepsen S, Pascual La Rocca A. Efficacy of professionally administered chemical agents as an adjunctive treatment to sub-marginal instrumentation during the therapy of peri-implant mucositis. J Clin Periodontol. 2023 Jun;50 Suppl 26:146-160. doi: 10.1111/jcpe.13747. Epub 2022 Dec 16. PMID 36375839
- [Background] Brunot-Gohin C, Duval JL, Azogui EE, Jannetta R, Pezron I, Laurent-Maquin D, Gangloff SC, Egles C. Soft tissue adhesion of polished versus glazed lithium disilicate ceramic for dental applications. Dent Mater. 2013 Sep;29(9):e205-12. doi: 10.1016/j.dental.2013.05.004. Epub 2013 Jun 24. PMID 23806786
- [Background] Blasi A, Iorio-Siciliano V, Pacenza C, Pomingi F, Matarasso S, Rasperini G. Biofilm removal from implants supported restoration using different instruments: a 6-month comparative multicenter clinical study. Clin Oral Implants Res. 2016 Feb;27(2):e68-73. doi: 10.1111/clr.12530. Epub 2014 Dec 11. PMID 25496020
- [Background] Barreto LAL, Grangeiro MTV, Prado PHCO, Bottino MA, Dal Piva AMO, Ramos NC, Tribst JPM, Junior LN. Effect of Finishing Protocols on the Surface Roughness and Fatigue Strength of a High-Translucent Zirconia. Int J Dent. 2023 Sep 22;2023:8882878. doi: 10.1155/2023/8882878. eCollection 2023. PMID 37780934